CLINICAL TRIAL: NCT03214393
Title: Role of Maternal Anticardiolipin and Anti-B2 Glycoprotein I Antibodies in Correlation With Fetal Doppler in Prediction of Adverse Pregnancy Outcome in Patients With Preeclampsia
Brief Title: Certain Maternal Antibodies in Relation to Doppler in Hypertension With Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Shafie Belal, Principal investigator, Cairo University
Other Study IDs: 3650
Record Dates: First submitted 2017-07-10; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-Eclampsia: pregnant women with Pre-Eclampsia will be assessed by serum antibodies and Doppler
  Interventions: Diagnostic Test: Doppler; Diagnostic Test: serum antibodies

INTERVENTIONS:
Diagnostic Test: Doppler — Doppler will be done to pregnant women with Pre-Eclampsia
Diagnostic Test: serum antibodies — serum antibodies will be measured for pregnant women with Pre-Eclampsia

SUMMARY:
Relation of certain maternal serum antibodies to Doppler changes will be studied in cases suffering from hypertension with pregnancy.

DETAILED DESCRIPTION:
Assessment will be done for maternal serum anti-beta 2 glycoprotein 1 antibodies and anticardiolipin antibodies in cases of preeclampsia after 32 weeks of pregnancy. In addition, fetal Doppler changes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 32 weeks or more gestational age
* Pre-eclampsia
* Singleton pregnancy

Exclusion Criteria:

* Intrauterine fetal death
* Fetus with apparent congenital anomalies
* Pregnant females with other medical disorders
* History of essential hypertension.
* History of antepartum hemorrhage.
* History of rupture of membranes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant females 32 weeks gestation or more with pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
percentage of cases that develop severe pre-eclampsia | It will be calculated after 1 year from the start of the study
  percentage of cases that develop severe pre-eclampsia will be assessed by an investigator

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Sh Belal, MD, Principal Investigator — Cairo U
Locations (1):
- Department of Obstetrics and Gynecology, Cairo, Greater Cairo, Egypt